CLINICAL TRIAL: NCT04442685
Title: The Swiss Registry for Heart Diseases in Children A Datacollection for Congenital and Acquired Heart Diseases in Children Living in Switzerland.
Brief Title: The Swiss Registry for Heart Diseases in Children Living in Switzerland. SPHC
Acronym: SPHC
Status: Completed | Type: Observational
Sponsor: University Children's Hospital, Zurich (Other)
Collaborators: Ostschweizer Kinderspital (Other); Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Christian Balmer, Principal Investigator Dr. Christian Balmer, University Children's Hospital, Zurich
Other Study IDs: BASEC 2018-01229
Record Dates: First submitted 2019-03-29; First posted 2020-06-22 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Heart Disease Congenital
Keywords: congenital heart disease; pediatric; registry; heart disease
MeSH Terms: conditions — Heart Defects, Congenital; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Swiss Pediatric Heart Cohort aims to collect representative longitudinal data on all children diagnosed with a clinically relevant heart disease in Switzerland. The long-term goal is to optimize diagnosis and therapy, and to allow setting up national research projects.

DETAILED DESCRIPTION:
In the entire spectrum of childhood diseases, heart disease occupy a special position regarding incidence; Congenital heart defects are among the most common organ abnormalities, moderate and severe forms of congenital heart diseases occur with a frequency of about 6 to 8 per 1000 live births. Rapid advances in diagnostic and therapeutic options in recent decades have led to a spectacular improvement in prognosis.

So far, data from heart diseases in children in Switzerland are not recorded centrally. A national registry collecting all relevant personal and medical data, as in other European countries, e.g. Finland, Sweden or Germany does not exist. The incidence and course of heart diseases in children in Switzerland are therefore unknown and can only be extrapolated indirectly from other countries. The SPHC project was therefore initiated by the Swiss pediatric cardiologists and is supported by its professional association, the Swiss Society for Pediatric Cardiology (Schweizerische Gesellschaft für pädiatrische Kardiologie; SGPK), as well as by its research association, the Association for Pediatric Heart Research Switzerland (Verein Kinderherzforschung Schweiz; VKHFS).

The aim of medical efforts in children with heart disease has shifted in recent years from a mere assurance of survival to an overall optimization of morbidity. These patients are expected to have a good perspective with normal growth, development, and quality of life well into adulthood. This goal can be achieved by researching the incidence and disease progression as well as the diagnostic and therapeutic measures in Switzerland. In this way, conclusions can be drawn, which lead to a modification of the therapeutic procedures and finally improve the prognosis of heart disease. The statistical significance of individual case descriptions or retrospective case series of individual centers, as practiced today, is insufficient for these purposes.

The aim of the SPHC is to optimize the diagnosis and therapy of all children with heart disease in Switzerland. In particular, the following goals are pursued:

* Describe incidence of heart diseases in childhood
* Enable research on the cause of the disease
* Record long-term history of mortality, morbidity and quality of life
* Describe therapeutic measures (medications, cardiac catheterization, cardiac surgery) regarding efficacy and safety
* Identify risk factors for a good / bad prognosis
* Promote prevention
* Collect basic data for the planning of care and for health economic analyses in the context of public health research projects
* Provide data for international collaborative studies
* A collaboration with Registry of adults with congenital heart defects (Grown Up Congenital Heart Disease, GUCH) is anticipated. This registry also uses SecuTrial® and is also located in the Clinical Trial Centre (CTC) of the University Zürich.

ELIGIBILITY:
Inclusion Criteria:

* Patients with heart diseases and
* age at diagnosis between 0 and 18 years and
* resident and / or treated in Switzerland and
* signed informed consent

Exclusion Criteria:

* No written consent. The number of people who refuse to participate will be recorded per center for drop out analysis.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The population from newborns to adolescents with newly diagnosed heart disease is recorded.
Sampling Method: Non-Probability Sample
Enrollment: 590 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
SPHC, a prospective quantitative datacollection of heart diseases in Swiss children during ten years. | Datacollection during 10 years, whereas an average incident is detected during one year
  This registry is a prospective data collection. It includes all patients who are newly diagnosed with a heart disease and who have consented to it. As the amount of data increases, the registry becomes more important and informative.
  The primarily outcome is to evaluate the quantity of congenital and acquired heart diseases in children living in Switzerland per Year compared to other countries.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Balmer, Principal Investigator — PI
Locations (1):
- University Childrens Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Specific research projects: At the request of researchers, the SPHC is used for focused research projects. For example, a questionnaire study to patients and their parents to assess quality of life and health, or a survey to attending physicians for detailed treatment modalities. The additional data gained in these projects will be fed back into the database.
  Networking: In the future there is a possibility that the data of the SPHC can be networked with further registries: e.g. Swiss Birth Registry (Swiss Federal Statistical Office), Swiss National Cohort, RADIZ: Registry for Rare Diseases, Swiss Ped Net and possible further registries. Also the cooperation with the registry for adults with congenital heart diseases (GUCH Registry) is essential and an inclusion of all SPHC patients reaching the age of 18 years in the GUCH registry is anticipated.
Supporting Information: Study Protocol
Time Frame: The first Data will be available 2020.
Access Criteria: all IPD that underlie results in a publication
URL: http://www.kinderherzforschung.ch

REFERENCES:
- See also: Prevalence of congenital heart defects — https://www.ncbi.nlm.nih.gov/pubmed/?term=Reller+MD%2C+Strickland+MJ%2C+Riehle-Colarusso+T%2C+Mahle+WT%2C+Correa+A.+Prevalence+of+congenital+heart+defects+in+metropolitan+Atlanta%2C+1998-2005.+J+Pediatr.+2008+Dec%3B153(6)%3A807-13.
- See also: Incidence of congenital heart defects — https://www.ncbi.nlm.nih.gov/pubmed/?term=Hoffman+JI%2C+Kaplan+S.+The+incidence+of+congenital+heart+disease.+Journal+of+the+American+College+of+Cardiology.+2002+Jun+19%3B39(12)%3A1890-900